CLINICAL TRIAL: NCT06317103
Title: A Retrospective, Single Center, Double Arm, Blind, Controlled, Pivotal Trial to Evaluate Classification by the Depth of Invasion of Early Gastric Cancer Sensitivity and Specificity of Gastric Cancer Image Computer Aided Detection and Diagnosis Software 'WAYMED Endo' and Endoscopists in Endoscopic Images
Brief Title: A Clinical Trial to Evaluate the Sensitivity and Specificity of "WAYMED Endo" Compared to the Endoscopists in Classifying Early Gastric Cancer (EGC) Based on the Depth of Invasion in Endoscopic Images
Status: Completed | Type: Observational
Sponsor: WAYCEN Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: WAY-CTP-WME01-MSM
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Early Gastric Cancer
Keywords: The depth of invasion categories for EGC (mucosal invasion, submucosal invasion)
MeSH Terms: conditions — Stomach Neoplasms | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trial group: The gastro-endoscopic images in this group are classified as "Mucosa" or "Submucosa" by WADYMED endo.
  Interventions: Device: WADYMED endo
- Control group: The gastro-endoscopic images in this group are interpreted as "Mucosa" or "Submucosa" by the endoscopists.
  Interventions: Other: Control group (the endoscopists)

INTERVENTIONS:
Device: WADYMED endo — Classification of the gastro-endoscopic images as "Mucosa" or "Submucosa" by WADYMED endo (Gastric cancer image, computer aided detection/diagnosis software)
  Groups: Trial group
Other: Control group (the endoscopists) — Interpretation of the gastro-endoscopic images as "Mucosa" or "Submucosa" by the endoscopists
  Groups: Control group

SUMMARY:
The purpose of this clinical trial is to prove that the prediction capability of 'WAYMED endo' is superior to that of the endoscopists in classifying EGC based on the depth of invasion categories in gastro-endoscopic images.

The computer-aided detection·diagnosis software is an Artificial Intelligence (AI) software used to assist medical specialists in diagnostic decisions by automatically classifying EGC based on the depth of invasion categories in gastro-endoscopic images and displaying the results and possibilities on the User Interface (UI).

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the sensitivity and specificity of 'WAYMED endo' compared to that of endoscopists in classifying EGC based on the depth of invasion categories in gastro-endoscopic images. It is designed as a retrospective, single-center, double-arm, double-blind (endoscopist, investigational medical device applicator), controlled, and pivotal trial. Medical data collected retrospectively from subjects who underwent Esophagogastroduodenoscopy (EGD) and biopsy are screened. As a result of screening, medical data that meet all inclusion/exclusion criteria are enrolled and assigned to the trial and control groups.

In the trial group, the investigational medical device is applied to the images, while the endoscopists interpret the images in the control group. The Reference Standard Establishment Committee records the reference standard results as either "Mucosa (mucosal invasion)" or "Submucosa (submucosal invasion)", based on the depth of invasion of the lesion, and marks the detected lesion area with an oval on the image. The reference standard results are blinded, so they cannot be disclosed to the endoscopists or the investigational medical device applicator.

The primary endpoint includes the sensitivity (%) and specificity (%) of "WAYMED endo" and the endoscopists in classifying EGC based on the depth of invasion categories ("Mucosa" or "Submucosa") as confirmed by the reference standard. The secondary endpoint includes the accuracy (%) of "WAYMED endo" and the endoscopists in accurately classifying all early gastric cancer images as either "Mucosa" or "Submucosa", based on the depth of invasion categories as confirmed through pathological examination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years or older who underwent EGD 2. Confirmed the presence of gastric cancer through the Electronic Medical Record (EMR), including reports of EGD or pathology

1. M ("Mucosa (mucosal invasion)"): Medical data of early gastric cancer patients with confirmed "Mucosa" for the depth of invasion category in the EMR.
2. SM ("Submucosa (submucosal invasion)"): Medical data of early gastric cancer patients with confirmed "Submucosa" for the depth of invasion category in the EMR.

Exclusion Criteria:

1. Absence of pathological results for the lesion
2. History of gastrectomy
3. Judged as inappropriate for inclusion by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastro-endoscopic images of early gastric cancer patients who underwent EGD
Sampling Method: Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Clinical Sensitivity in classifying early gastric cancer (EGC) based on the depth of invasion (%) | 3 months
  The probability of being classified as "Mucosa (mucosal invasion)", based on the depth of invasion categories for early gastric cancer, among gastro-endoscopic images confirmed as "Mucosa" through the results of pathologic examination.
Clinical Specificity in classifying early gastric cancer (EGC) based on the depth of invasion (%) | 3 months
  The probability of being classified as "Submucosa (submucosal invasion)", based on the depth of invasion categories for early gastric cancer, among gastro-endoscopic images confirmed as "Submucosa" through the results of pathologic examination.

SECONDARY OUTCOMES:
Accuracy in classifying the depth of invasion categories ("Mucosa" or "Submucosa") for early gastric cancer (%) | 3 months
  The probability of accurately classifying all early gastric cancer images as either "Mucosa" or "Submucosa", based on the depth of invasion categories confirmed through pathological examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jie-Hyun Kim, Principal Investigator — Yonsei University Gangnam Severance Hospital
Locations (1):
- Yonsei University Gangnam Severance Hospital, Seoul, South Korea